CLINICAL TRIAL: NCT01633125
Title: Group Music Therapy for Chinese Prisoners: A Randomized Controlled Trial
Brief Title: Group Music Therapy for Chinese Prisoners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Xi Jing Chen, Cand. PhD, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aau-1
Record Dates: First submitted 2012-06-25; First posted 2012-07-04 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-06

CONDITIONS: Anxiety; Depression; Self-esteem
Keywords: Group music therapy; prisoners; Anxiety; Depression; Self-esteem
MeSH Terms: conditions — Anxiety Disorders; Depression

ARMS (2):
- Group music therapy (Experimental): Participants in the experimental group will take part in biweekly group music therapy for 10 weeks (20 sessions). Each group will be formed by 6 to 8 people, and each session will last for 90 minutes.The academically trained music therapist with previous relevant clinical experience will apply receptive and active music therapy techniques. The active techniques will include musical improvisation as a medium to work with participants according to therapeutic goals and participants' needs.
  Interventions: Other: Group music therapy
- No music therapy (No Intervention): Participants assigned to the control group will not receive any specific treatment in this study. The usual care that is normally available at the prison will continue to be available for all participants during the study.Due to ethical considerations, the control group will receive group music therapy or psychotherapy by academically qualified therapists for 5 weeks after the study is finished.
  Interventions: Other: Group music therapy

INTERVENTIONS:
Other: Group music therapy — The academically trained music therapist with previous relevant clinical experience will apply receptive and active music therapy techniques. The receptive methods will include music imagery,The active techniques will include musical improvisation and song writing.
  Other Names: Music imagery; Song writing; Improvisation

SUMMARY:
The prevalence of psychological problems is high in prisons. Many prisoners have unmet needs for appropriate treatments. Although pilot studies have suggested music therapy to be a successful treatment modality for prisoners, more rigorous evidence is needed.

This study aims to investigate the effectiveness of group music therapy to improve anxiety, depression, and self-esteem in prisoners. One hundred and ninety two inmates from a Chinese prison will be allocated to two groups through randomisation. The experimental group will participate in biweekly group music therapy for 10 weeks (20 sessions) while the control group will be placed on a waitlist. Anxiety, depression and self-esteem will be measured by self-report scales three times: before, at the middle, and at the end of the intervention. Logs by prisoners and daily behavior observation by trained prison guards will be used as additional information.

This study will increase the knowledge of the effectiveness of group music therapy. Results will be generalizable to Chinese prisons but also internationally. Generalizability to clinical practice will be high, and findings will be able support the further development of music therapy in prison.

DETAILED DESCRIPTION:
Objectives

* The purpose of this study is to examine the effectiveness of group music therapy in prison. Specifically, the investigators aim to determine whether group music therapy is associated with greater improvements in levels of anxiety, depression, and self-esteem among prisoners than the care that is normally provided. Additionally the investigators aim to explore the unique value of music therapy in prison, its potential advantages to other forms of therapy in this setting, and how it can be effectively implemented in the Chinese prison system.

Methods

* A randomized controlled study with individual assignment of participants to one of two parallel groups will be conducted to determine the effects of group music therapy compared to no treatment.

Participants

* Inmates from a prison in Beijing, China will be eligible to participate in this study and will be included if they are willing and meet the inclusion criteria detailed below. Recruitment started in April 2012 and will continue until 192 participants have been enrolled during this period.

Interventions

* Experimental group

  * Participants in the experimental group will take part in biweekly group music therapy for 10 weeks (20 sessions). Each group will be formed by 6 to 8 people, and each session will last for 90 minutes. The sessions will take place in the activity room in the prison. The academically trained music therapist with previous relevant clinical experience will apply receptive and active music therapy techniques. The active techniques will include musical improvisation as a medium to work with participants according to therapeutic goals and participants' needs. The music therapist has a background in both psychodynamic and humanistic approaches, but will apply existential-humanistic oriented approaches to work with the participants of this study. Taking into account factors such as the limited duration of the intervention, the outcomes of this study, and the group setting of the intervention, the humanistic framework is felt to be more suitable for this study than a psychodynamic framework. Specifically, the outcomes including emotions and self-esteem are closely related to the humanistic approach. The therapist will focus on creating a favorable and respectful environment, building trustful and authentic relationships between the therapist and group members, and increasing their self-awareness, encouraging the participants' expression and sharing of emotions.

The first three sessions will be introductory sessions. The music therapist will introduce the goals of music therapy, three techniques of music therapy (improvisation, song writing, and music imagery), and discuss how these approaches can help the group. Each the following session will start with a discussion on the focus of the group (the thoughts, emotions, or topics which the group wants to share or explore). Then, the therapist and the group will reach an agreement which music therapy technique should be chosen. The therapist will keep the flexibility of music therapy techniques applied in this study to ensure the result of this research to be closely related to clinical work. In usual clinical work, music therapists tend to apply multiple methods in working with clients. At the end of each session, the group members will reflect on the music therapy activity through verbal discussion, drawing, or other musical experiences (such as another improvisation, singing a song together, or movement in music) to bring the session to a closure.

* Control group

  * Participants assigned to the control group will not receive any specific treatment in this study. The usual care that is normally available at the prison will continue to be available for all participants during the study. This may include medical care and psychological/psychotherapeutic care. The rate of psychotherapy is usually very low, except in case of any extreme events (such as suicidal behavior, severe outbursts of anger, or fights with other prisoners). All prisoners will normally have a psychological class together. Data will be collected of how many participants in each group received other therapies during the study. Due to ethical considerations, the control group will receive group music therapy or psychotherapy by academically qualified therapists for 5 weeks after the study is finished.

Study Design

The investigators will allocate participants individually to the interventions using a computer-generated randomization list. Randomization will be balanced within prison departments to ensure equal sizes of intervention groups. This will not compromise allocation concealment because eligible participants from one department will be randomized simultaneously (rather than entering the study successively one by one). A person who has no direct contact with participants will conduct the randomization so that concealment of allocation can be assured before the intervention.

Because of the scarcity of qualified music therapists in Chinese prisons, the first author will also be the music therapist to execute intervention. An advantage of this double role may be that this experience will allow her to be closely involved in the therapy process and to closely observe and experience changes in the participants. This vivid process will facilitate the interpretation of the data because it will help to understand any unexpected results through the therapist's experience and observation from the music therapy sessions. The quality of the therapy will be ensured through weekly supervision with an experienced music therapist. A qualified psychotherapist will be trained to help the participants to complete the self-report scales. This person will ensure that participants understand the questions and complete the questionnaire correctly, but will not be involved in the therapy and will be instructed not to influence the participants in their ratings. The behavioral observations will be collected by the prison guards who will be unaware of the purpose of this study.

Outcomes of this study will be assessed at pre-test (before randomization; these measurements will also be used to screen participants), at the mid-point of the intervention (after 5 weeks) and at post-test (after 10 weeks). A longer follow up investigation is not possible because participants in the control group will be offered therapy after post-test.

ELIGIBILITY:
Inclusion Criteria:

* Without diagnosis of psychotic problems
* Show a higher level of anxiety or depression level than the average level of the normal population.
* Have a remaining sentence of 6 months or more from the date of enrollment into the study.

Exclusion Criteria:

* With severe physical diseases
* With psychotic disorders
* Intelligence quotient is ≤69 (mild mental retardation)
* Unable to understand and complete the questionnaires

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in State Trait Anxiety Inventory at 10 weeks | Baseline and 10 weeks
  Anxiety will be measured with the State Trait Anxiety Inventory (STAI). The STAI contains two subscales that are relatively similar, and a qualified person will be present to make sure the participants understand the difference between them. The first subscale measures state anxiety (reflecting the current level of anxiety which can change quickly), whereas the second measures trait anxiety (reflecting anxiety as a more general trait that may also change over time but is more lasting than state anxiety).
Change from baseline in State Trait Anxiety Inventory at 20 weeks | Baseline and 20 weeks

SECONDARY OUTCOMES:
Change from baseline in Beck Depression Inventory at 10 weeks | Baseline and 10 weeks
  Depression will be assessed using the Beck Depression Inventory (BDI). This instrument consists of 21 items; the score of each item ranges from 0 to 3, producing a total range from 0 to 63, with higher scores indicating greater depression. BDI has become one of the most widely used instruments not only for assessing the intensity of depression in psychiatric patients, but also for detecting depression in normal populations.
Change from baseline in Beck Depression Inventory at 20 weeks | Baseline and 20 weeks
Change from baseline in Rosenberg Self-esteem Inventory at 10 weeks | Baseline and 10 weeks
  Self-esteem will be assessed as a secondary outcome. It will be assessed using two self-report scales, the Rosenberg Self-esteem Inventory (RSI) and the Texas Social Behavior Inventory (TSBI). RSI and TSBI measure global self-esteem and social self-esteem, respectively.
Change from baseline in Rosenberg Self-esteem Inventory at 20 weeks | Baseline and 20 weeks
Change from baseline in Texas Social Behavior Inventory at 10 weeks | Baseline and 10 weeks
  Self-esteem will also be assessed as a secondary outcome. It will be assessed using two self-report scales, the Rosenberg Self-esteem Inventory (RSI) and the Texas Social Behavior Inventory (TSBI). RSI and TSBI measure global self-esteem and social self-esteem, respectively.
Change from baseline in Texas Social Behavior Inventory at 20 weeks | Baseline and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jing X Chen, Master, Principal Investigator — Aalborg University
Locations (1):
- Xin An Prison, Beijing, Beijing Municipality, China